CLINICAL TRIAL: NCT07291440
Title: Impact of Balneotherapy in Ma'n Hot Spring on Quality of Life in Adult With Low Back Pain: Randomized Clinical Trial
Brief Title: Impact of Balneotherapy in Ma'n Hot Spring on Quality of Life in Adults With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Kerolous Ishak Shehata, Lecturer at physical therapy department for women's health, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#27\9\2025-2026
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain
Keywords: Ma'n hot spring; quality of life; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): The study group will perform regular aerobic exercise on mat
  Interventions: Other: Core stability exercise
- Ma'n hot spring (Experimental): The experimental group will perform underwater exercise in Ma'n hot spring
  Interventions: Other: Core stability exercise

INTERVENTIONS:
Other: Core stability exercise — The core is a box structure made up of the abdominal muscles in the front and the sides, the paraspinal and gluteal muscles at the back, the diaphragm at the roof, and the pelvic floor and the hip girdle muscles as the floor.

SUMMARY:
Effect of Ma'n hot spring on quality of life in adults with low back pain

DETAILED DESCRIPTION:
Effect of Ma'n hot spring on quality of life in adults with low back pain

ELIGIBILITY:
Inclusion Criteria:

* BMI> 25
* low muscle power
* low quality of life
* general fatigue

Exclusion Criteria:

* BMI< 25
* Polycystic ovarian syndrome
* Chronic pelvic pain
* Lumbar disc

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Biofeedback | Start before starting aerobic exercise and after 6 weeks of performing 12 sessions
  Biofeedback is a valuable tool for assessing and training muscle power in the lower back region. It involves using pressure biofeedback units to measure the strength of core muscles such as the transversus abdominis and lumbar multifidi. Pressure ranged from zero to 100 and zero point means weak muscle and 100 means high power muscle
Visual analogue scale | Before starting aerobic exercise and after 6 weeks of performing 12 sessions
  It is a scale ranged from zero to ten and zero point indicate there is no pain and ten point indicate the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Kerolous IS Kelini, Principal Investigator — Al-Zaytoonah University
Locations (1):
- AL-Zaytoonah University, Amman, Jordan